CLINICAL TRIAL: NCT05376852
Title: Decitabine and HQP1351-based Chemotherapy Regimen for the Treatment Advanced Chronic Myeloid Leukemia
Brief Title: Decitabine and HQP1351-based Chemotherapy Regimen for the Treatment Advanced CML
Acronym: Case-Only
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xuna, professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML220520
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Chronic Myeloid Leukemia in Myeloid Blast Crisis; Chronic Myeloid Leukaemia Transformation; Chronic Myeloid Leukemia - Accelerated Phase; Chronic Myeloid Leukemia in Lymphoid Blast Crisis
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Based decitabine and olverembatinib（HQP1351)chemotherapy
  Interventions: Combination Product: based decitabine and olverembatinib（HQP1351)chemotherapy

INTERVENTIONS:
Combination Product: based decitabine and olverembatinib（HQP1351)chemotherapy — AP-CML treated with decitabine 10mg/m2 d1-5 intravenously (IV) over 60 minutes on days 1-5 and HQP1351 40mg qod every 28 days.After completion of HQP1351 lead-in, patients will receive HQP1351 PO qod on days 1-28 of subsequent cycles.
  BC-CML:treated with decitabine 20mg/m2 d1-5 IV on days 1-5 and HQP1351 40mg qod every 28 days,with or without other chemotherapy Drugs

SUMMARY:
This phase II trial studies how well the combination of based decitabine and olverembatinib（HQP1351)chemotherapy work for the treatment of blast phase or accelerated phase chronic myelogenous leukemia. Drugs used in chemotherapy such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. HQP1351 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving decitabine and ponatinib based chemotherapy may help to control blast phase or accelerated phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
Accelerated Phase CML treated with decitabine10mg/m2 d1-5 intravenously (IV) over 60 minutes on days 1-5 and olverembatinib（HQP1351) 40mg qod every 28 days.After completion of HQP1351 lead-in, patients will receive HQP1351 PO daily on days 1-28 of subsequent cycles.

chronic myeloid leukaemia in blast phase:treated with decitabine 20mg/m2 d1-5 intravenously (IV) over 60 minutes on days 1-5 and HQP1351 40mg qod every 28 days,with or without other chemotherapy drugs

ELIGIBILITY:
Inclusion Criteria:

* myeloid accelerated phase (AP)-chronic myelogenous leukemia (CML) or blast phase (BP)-CML (either t[9;22] and/or BCR-ABL1 positive by fluorescent in situ hybridization or polymerase chain reaction). Both untreated and relapsed/refractory patients are eligible
* Performance status =< 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 2 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the principal investigator (PI) Alanine aminotransferase (ALT) =< 1.5 x ULN, unless due to the underlying leukemia approved by the PI Aspartate aminotransferase (AST) =< 1.5 x ULN unless due to the underlying leukemia approved by the PI Creatinine clearance >= 30 mL/min Serum lipase =< 1.5 x ULN Amylase =< 1.5 x ULN Ability to swallow Signed informed consent

Exclusion Criteria:

Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment) History of acute pancreatitis within 6 months of study or history of chronic pancreatitis Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL) Active secondary malignancy that in the investigator's opinion will shorten survival to less than 1 year Active grade III-V cardiac failure as defined by the New York Heart Association criteria

Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

Myocardial infarction (MI), stroke, revascularization, unstable angina or transient ischemic attack within 6 months Left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards prior to enrollment Diagnosed or suspected congenital long QT syndrome Clinically significant atrial or ventricular arrhythmias (such as uncontrolled, clinically significant atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes) as determined by the treating physician Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 480 msec) unless corrected after electrolyte replacement History of venous thromboembolism including deep venous thrombosis or pulmonary embolism within the past 3 months, excluding line-associated deep venous thrombosis (DVT) of the upper extremity Uncontrolled hypertension (diastolic blood pressure > 100 mmHg; systolic > 150 mmHg)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At 12 weeks
  Defined as the proportion of patients achieving complete remission (CR) + CR with incomplete count recovery (CRi) occurring at the end of 2 cycles of treatment. Will be estimated along with the 95% credible interval. Patients who drop out of the study before completing 2 cycles and have been treated will be censored for the primary endpoint analysis.

SECONDARY OUTCOMES:
Relapse-free survival | 3 years
  From documented complete response until relapse or death
Event-free survival | 3 years
  From first day of treatment until any failure (resistant disease, relapse, or death)
Overall survival | assessed up to 3 years
  First day of treatment to time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Nanfang Hospital, Southern Medical University,, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No